CLINICAL TRIAL: NCT02113358
Title: Comparison of Stroke Volume Variation-guided Normovolemic and Restrictive Fluid Management During Craniotomy: a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201312116RINC
Record Dates: First submitted 2014-04-08; First posted 2014-04-14 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Supratentorial Neoplasms; Brain Tumor, Primary; Craniotomy
Keywords: fluid therapy; neurosurgery
MeSH Terms: conditions — Supratentorial Neoplasms; Brain Neoplasms | interventions — HES 130-0.4

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normovolemic group (keeping SVV<10% in supine; <15% in prone) (Experimental): 1. The anesthesiologist will infuse Voluven (Fresenius Kabi, Bad Homburg, Germany) 250 ml if stroke volume variation is over 10% during the surgery to keep the normovolemia.
  2. If total Voluven use is over 1500ml and then the anesthesiologist will infuse Saline 250 ml instead.
  3. The maintenance of basal fluid, criteria to use inotropes (If cardiac index is below 2.5 l/min/m2 ) are the same standards in the both groups.
  Interventions: Drug: Intravenous colloid bolus with Voluven
- Restricitve group (keeping SVV < 18% in supine; <23% in prone) (Active Comparator): 1. The anesthesiologist will infuse Voluven (Fresenius Kabi, Bad Homburg, Germany) 250 ml if stroke volume variation is over 18% during the surgery to keep the normovolemia.
  2. If total Voluven use is over 1500ml and then the anesthesiologist will infuse Saline 250 ml instead.
  3. The maintenance of basal fluid, criteria to use inotropes (If cardiac index is below 2.5 l/min/m2 ) are the same standards in the both groups.
  Interventions: Drug: Intravenous colloid bolus with Voluven

INTERVENTIONS:
Drug: Intravenous colloid bolus with Voluven

SUMMARY:
Fluid management during neurosurgery presents a special clinical agenda. Volume overload can have detrimental effects on intracranial pressure by increasing either cerebral blood volume or hydrostatically driven cerebral edema formation. On the other hand, an overt restrictive fluid strategy may risk hemodynamic instability.

Recently, dynamic fluid responsiveness parameters such as stroke volume variation (SVV) have been shown as a more precise parameters for fluid management including in neurosurgical patients. The threshold of SVV is reported about 10-15%. In this study, the investigators aim to using two SVV threshold to conduct intraoperative fluid therapy for craniotomy. Randomization will be generated by computer sampling. One of the two groups of patients will be managed with fluid bolus to keep intraoperative SVV <10% presenting the "normovolemia" group. The other group of patients will be kept intraoperative SVV <18% which is slightly above previously reported SVV threshold upper limit. The second group thus presents the "restrictive" group. Clinical outcomes, laboratory analysis including S100-B for neuronal damage and neutrophil gelatinase-associated lipocalin (NGAL) for acute kidney injury, will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Supratentorial brain tumor receiving elective craniotomy
* BMI between 18.5-27.0 kg.m-2

Exclusion Criteria:

* Cardiac dysfunction, such as coronary artery diseases; atrial fibrillation;

  * NYHA class II
* Renal dysfunction, eGFR< 60 ml.min-1.1.73m-2
* Pulmonary cormorbidity, such as COPD

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
serum S100B protein | Changes from preoperative to postoperative day 2
serum NGAL level | Changes from preoperative to postoperative day 2.

SECONDARY OUTCOMES:
Length of hospital stay | participants will be followed for the duration of hospital stay, an expected average of 3 to 4 weeks
Postoperative complications rate | participants will be followed for the duration of hospital stay, an expected average of 3 to 4 weeks
Total intraoperative intravenous fluid administrated | During the surgical time, an expected average of 3 to 5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Yu Wu, MD, Principal Investigator — National Taiwan University Hospital Anesthesiology Department
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Wu CY, Lin YS, Tseng HM, Cheng HL, Lee TS, Lin PL, Chou WH, Cheng YJ. Comparison of two stroke volume variation-based goal-directed fluid therapies for supratentorial brain tumour resection: a randomized controlled trial. Br J Anaesth. 2017 Nov 1;119(5):934-942. doi: 10.1093/bja/aex189. PMID 28981592